CLINICAL TRIAL: NCT01306292
Title: A Phase II, Double-Blind, Randomized, Placebo-Controlled, Crossover, Safety Study of the Effect of Intravenous Bolus Injections of SonoVue on Pulmonary Hemodynamics in Subjects With and Without Pulmonary Hypertension
Brief Title: Safety of SonoVue on Pulmonary Hemodynamics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: BR1-133
Record Dates: First submitted 2011-02-23; First posted 2011-03-01 (Estimated); Results first posted 2016-02-08 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-10

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary hypertension; Right heart Catheterization
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — contrast agent BR1; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SonoVue (Experimental): Ultrasound contrast agent under development
  Interventions: Drug: SonoVue
- Placebo (Placebo Comparator): normal saline 0.9% for injection used as the comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SonoVue — dose of 4.8 mL administered intravenously one time
  Other Names: sulfur hexafluoride microbubbles; sulfur hexafluoride lipid-type A microspheres
  Arms: SonoVue
Drug: Placebo — Placebo is normal saline 0.9% for injection used as the comparator administered at 4.8 mL (same dose as SonoVue)
  Other Names: Normal Saline
  Arms: Placebo

SUMMARY:
This is an intra-subject crossover comparative safety study to evaluate the effect of intravenous (IV) bolus injection of SonoVue on pulmonary hemodynamics.

DETAILED DESCRIPTION:
Subjects will be divided into two groups based on their baseline mean pulmonary arterial pressure. Each subject will receive two injections in randomized order during right heart catheterization: one administration of SonoVue and one administration of placebo, either SonoVue followed by Placebo or Placebo followed by SonoVue. The purpose is to provide direct evidence on the presence or absence of pulmonary hemodynamic effect following IV administration of SonoVue versus any effects following IV administration of the same volume of placebo.

ELIGIBILITY:
Inclusion Criteria:

* Provides written informed consent male or female at least 18 years of age scheduled to undergo right heart catheterization for clinical reasons

Exclusion Criteria:

* Pregnant or lactating females
* Significant arrhythmia or non-sinus rhythm that may affect the ability to assess pulmonary hemodynamics by catheterization
* Known allergy to one of the ingredients in the investigational product or to any other contrast agents including ultrasound contrast agents
* Previously entered into the study or received an investigational compound within 30 days before admission into the study
* Unstable pulmonary and/or systemic hemodynamic condition that would affect the ability to evaluate the pharmacological or hemodynamic effect of the investigational products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-04; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Luigia Storto, MD, Study Director — Bracco Diagnostics, Inc
Locations (1):
- Holy Name Medical Center, Teaneck, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Study of Lumason pulmonary hemodynamics

RESULTS

PARTICIPANT FLOW:
Groups:
- Hypertension Group (SonoVue First, Then Placebo): Subjects with pulmonary hypertension (baseline mean pulmonary arterial pressure ≥ 25.0 mmHg) who were randomized to receive SonoVue first, then Placebo (normal saline 0.9% for injection). Both agents were administered intravenously as a single bolus injection of 4.8 mL. The two injection were separated by an interval of at least 10 minutes.
- Hypertension Group (Placebo First, Then SonoVue): Subjects with pulmonary hypertension (baseline mean pulmonary arterial pressure ≥25.0 mmHg) who were randomized to receive Placebo (normal saline 0.9% for injection) first, then SonoVue. Both agents were administered intravenously as a single bolus injection of 4.8 mL. The two injection were separated by an interval of at least 10 minutes.
- Normal Group (SonoVue First, Then Placebo): Subjects without pulmonary hypertension (baseline mean pulmonary arterial pressure <25.0 mmHg) who were randomized to receive SonoVue first, then Placebo (normal saline 0.9% for injection). Both agents were administered intravenously as a single bolus injection of 4.8 mL. The two injection were separated by an interval of at least 10 minutes.
- Normal Group (Placebo First, Then SonoVue): Subjects without pulmonary hypertension (baseline mean pulmonary arterial pressure <25.0 mmHg) who were randomized to receive Placebo (normal saline 0.9% for injection) first, then SonoVue. Both agents were administered intravenously as a single bolus injection of 4.8 mL. The two injection were separated by an interval of at least 10 minutes.
Period: First Injection
Arm/Group | Hypertension Group (SonoVue First, Then Placebo) | Hypertension Group (Placebo First, Then SonoVue) | Normal Group (SonoVue First, Then Placebo) | Normal Group (Placebo First, Then SonoVue)
Started | 10 | 8 | 8 | 10
Completed | 10 | 8 | 8 | 10
Not Completed | 0 | 0 | 0 | 0
Period: Washout (at Least 10 Minutes)
Arm/Group | Hypertension Group (SonoVue First, Then Placebo) | Hypertension Group (Placebo First, Then SonoVue) | Normal Group (SonoVue First, Then Placebo) | Normal Group (Placebo First, Then SonoVue)
Started | 10 | 8 | 8 | 10
Completed | 10 | 8 | 8 | 10
Not Completed | 0 | 0 | 0 | 0
Period: Second Injection
Arm/Group | Hypertension Group (SonoVue First, Then Placebo) | Hypertension Group (Placebo First, Then SonoVue) | Normal Group (SonoVue First, Then Placebo) | Normal Group (Placebo First, Then SonoVue)
Started | 10 | 8 | 8 | 10
Completed | 10 | 8 | 7 (1 subject completed both injections but not 24-hour follow-up; all other values were recorded.) | 10
Not Completed | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Hypertension Group: Subjects with pulmonary hypertension (baseline mean pulmonary arterial pressure ≥25.0 mmHg) who received SonoVue and Placebo (normal saline 0.9% for injection) in randomized order, both administered intravenously as a single bolus injection of 4.8 mL.
- Normal Group: Subjects without pulmonary hypertension (baseline mean pulmonary arterial pressure <25.0 mmHg) who received SonoVue and Placebo (normal saline 0.9% for injection) in randomized order, both administered intravenously as a single bolus injection of 4.8 mL.
- Total: Total of all reporting groups
Arm/Group | Hypertension Group | Normal Group | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 14 | 26
  >=65 years | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (12.96) | 57.2 (10.70) | 57.6 (11.72)
Gender [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 13 | 12 | 25
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Effects of SonoVue and Placebo on Pulmonary Hemodynamics: Systolic Pulmonary Artery Pressure (mmHg) - Mean Change From Baseline
Description: A total of 36 subjects were enrolled in this crossover study: 18 (8 randomized to placebo then SonoVue and 10 randomized to SonoVue then placebo) in the Hypertension Group (baseline mean pulmonary artery pressure (PAP) >=25.0 mmHg group) and 18 (10 randomized to placebo then SonoVue and 8 randomized to SonoVue then placebo) in the Normal group (baseline mean PAP <25.0 mmHg group). All subjects in this study were to have systolic PAP recorded within 5 minutes before the first investigational product administration. This parameter was to be measured and recorded again at 1, 4, 7 and 10 minutes after the administration of each investigational product (SonoVue and Placebo). This outcome measure presents the mean change from baseline in systolic PAP measured in mmHg. Baseline is the average of the 2 measurements within 5 minutes prior to first investigational product administration, therefore, applying to both products.
Time Frame: Comparison to baseline to 4 post dose timepoints (1, 4, 7 and 10 minutes post dose)
Population: 36 total subjects: 18 subjects (8 assigned to placebo/SonoVue and 10 assigned to SonoVue/placebo) in the Baseline mean PAP >=25.0 mmHg group (Hypertension Group) and 18 subjects (10 assigned to placebo/SonoVue and 8 assigned to SonoVue/placebo) in the Baseline mean PAP <25.0 mmHg group (Normal Group).
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Hypertension Placebo: Subjects with pulmonary hypertension (baseline mean pulmonary arterial pressure ≥ 25.0 mmHg) who received Placebo (normal saline 0.9%) administered intravenously as a single bolus injection of 4.8 mL.
- Hypertension SonoVue: Subjects with pulmonary hypertension (baseline mean pulmonary arterial pressure ≥ 25.0 mmHg) who received SonoVue administered intravenously as a single bolus injection of 4.8 mL.
- Normal Placebo: Subjects without pulmonary hypertension (baseline mean pulmonary arterial pressure < 25.0 mmHg) who received Placebo (normal saline 0.9%) administered intravenously as a single bolus injection of 4.8 mL.
- Normal SonoVue: Subjects without pulmonary hypertension (baseline mean pulmonary arterial pressure < 25.0 mmHg) who received SonoVue administered intravenously as a single bolus injection of 4.8 mL.
Arm/Group | Hypertension Placebo | Hypertension SonoVue | Normal Placebo | Normal SonoVue
Number analyzed (Participants) | 18 | 18 | 18 | 18
mmHg
  Baseline Systolic PAP (mmHg) | 50.50 (17.581) | 50.50 (17.581) | 30.08 (6.001) | 30.08 (6.001)
  1 minute post-dose | -2.17 (5.993) | -3.33 (5.407) | 1.31 (3.214) | 0.47 (2.464)
  4 minutes post-dose | -3.06 (5.196) | -2.94 (5.352) | 1.50 (4.345) | 0.62 (2.485)
  7 minutes post-dose | -1.94 (6.010) | -2.28 (4.854) | 0.86 (3.940) | -0.32 (2.215)
  10 minutes post-dose | -2.44 (6.849) | -2.17 (5.300) | 0.03 (4.816) | -0.69 (3.945)

2. Primary Outcome: Effects of SonoVue and Placebo on Pulmonary Hemodynamics: Diastolic Pulmonary Artery Pressure (mmHg) - Mean Change From Baseline
Description: All subjects in this study were to have diastolic PAP recorded within 5 minutes before the first investigational product administration. This parameter was to be measured and recorded again at 1, 4, 7 and 10 minutes after the administration of each investigational product (SonoVue and Placebo). This outcome measure presents the mean change from baseline in diastolic PAP measured in mmHg. Baseline is the average of the 2 measurements within 5 minutes prior to first investigational product administration, therefore, applying to both products.
Time Frame: Comparison to baseline to 4 post dose timepoints (1, 4, 7 and 10 minutes post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Hypertension Placebo | Hypertension SonoVue | Normal Placebo | Normal SonoVue
Number analyzed (Participants) | 18 | 18 | 18 | 18
mmHg
  Baseline Diastolic PAP (mmHg) | 24.11 (7.177) | 24.11 (7.177) | 11.72 (3.750) | 11.72 (3.750)
  1 minute post-dose | -3.39 (4.661) | -1.50 (3.884) | 1.44 (3.481) | 1.22 (4.156)
  4 minutes post-dose | -3.56 (4.362) | -2.78 (6.839) | 0.44 (3.508) | 0.68 (2.767)
  7 minutes post-dose | -3.22 (5.342) | -3.06 (4.325) | 1.61 (2.471) | 1.09 (3.104)
  10 minutes post-dose | -3.44 (5.731) | -1.83 (4.836) | 1.39 (2.207) | 0.78 (3.723)

3. Primary Outcome: Effects of SonoVue and Placebo on Pulmonary Hemodynamics: Pulmonary Vascular Resistance (Dyne*Sec/cm^5) - Mean Change From Baseline
Description: All subjects in this study were to have pulmonary vascular resistance (PVR; measured in dyne x seconds per centimeters to the 5th power) derived from mean PAP (measured in mmHg), pulmonary capillary wedge pressure (PCWP [mmHg]) and cardiac output (Qp [litres per minute]), each taken 5 minutes prior to the first investigational product administration, calculated using the following formula: [(mean PAP-PCWP) divided by Qp] x 80. Baseline is the last measurement prior to first investigational product administration, therefore, applying to both products. Mean PAP, PCWP and Qp were repeated at 1 and 10 minutes post dose; PVR was calculated.
Time Frame: Comparison to baseline to 2 post dose timepoints (1 and 10 minutes post dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: dyne*sec/cm^5
Arm/Group | Hypertension Placebo | Hypertension SonoVue | Normal Placebo | Normal SonoVue
Number analyzed (Participants) | 18 | 18 | 18 | 18
dyne*sec/cm^5
  Baseline PVR (dyne*sec/cm^5) | 307.189 (307.6268) | 307.189 (307.6268) | 142.714 (93.6055) | 142.714 (93.6055)
  1 minute post-dose | -73.087 (186.9939) | -63.065 (158.7097) | 20.541 (63.4305) | 1.021 (55.5296)
  10 minutes post-dose | -41.468 (226.7863) | -10.028 (175.0397) | 21.208 (82.9967) | -6.117 (52.0617)

ADVERSE EVENTS:
Time Frame: Adverse events were to be monitored from the time of signed informed consent until 24 hours after the last investigational product administration.
Groups:
- Hypertension Group: Subjects with pulmonary hypertension (baseline mean pulmonary arterial pressure ≥25.0 mmHg) who received SonoVue and Placebo (normal saline 0.9% for injection) in randomized order, both administered intravenously as a single bolus injection of 4.8 mL. An interval of at least 10 minutes was allowed between the two injections (SonoVue and Placebo). All adverse events occurred hours after the completion of both injections and for the purposes of this study have been assigned to the administration of SonoVue.
- Normal Pulmonary Pressure Group: Subjects without pulmonary hypertension (baseline mean pulmonary arterial pressure <25.0 mmHg) who received SonoVue and Placebo (normal saline 0.9% for injection) in randomized order, both administered intravenously as a single bolus injection of 4.8 mL. An interval of at least 10 minutes was allowed between the two injections (SonoVue and Placebo). All adverse events occurred hours after the completion of both injections and for the purposes of this study have been assigned to the administration of SonoVue.
Arm/Group | Hypertension Group | Normal Pulmonary Pressure Group
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 1/18 | 2/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hypertension Group (N=18) | Normal Pulmonary Pressure Group (N=18)
Catheter site pain (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days